CLINICAL TRIAL: NCT00497497
Title: A Phase Ib, Dose-Escalation Study of the Safety and Pharmacokinetics of PRO95780 in Combination With Cetuximab and Irinotecan Chemotherapy or the FOLFIRI Regimen With Bevacizumab in Patients With Previously Treated Metastatic Colorectal Cancer
Brief Title: A Study of PRO95780 in Combination With Cetuximab and Irinotecan Chemotherapy or the FOLFIRI Regimen With Bevacizumab in Patients With Previously Treated Metastatic Colorectal Cancer (APM4187g)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: APM4187g
Record Dates: First submitted 2007-07-03; First posted 2007-07-06 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Cancer
Keywords: CRC; Colon cancer; Avastin; APM4187g
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Bevacizumab; Cetuximab; Irinotecan; drozitumab

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: cetuximab; Drug: irinotecan; Drug: PRO95780
- 2 (Experimental)
  Interventions: Drug: bevacizumab; Drug: FOLFIRI regimen; Drug: PRO95780

INTERVENTIONS:
Drug: bevacizumab — (Only for patients not previously treated with bevacizumab) Intravenous repeating dose
  Arms: 2
Drug: cetuximab — Intravenous repeating dose
  Arms: 1
Drug: FOLFIRI regimen — Intravenous repeating dose
  Arms: 2
Drug: irinotecan — Intravenous repeating dose
  Arms: 1
Drug: PRO95780 — Intravenous repeating dose

SUMMARY:
This is a Phase Ib, open-label, multicenter, dose-escalation study designed to assess if PRO95780 in combination with two different irinotecan-containing regimens is safe and tolerable in patients with metastatic colorectal cancer (mCRC) who have progressed following, or cannot tolerate, first-line therapy with 5-fluorouracil-, oxaliplatin-, and bevacizumab-containing regimens. This study will also make a preliminary assessment of the anti-tumor activity of PRO95780 in combination with irinotecan and cetuximab or the FOLFIRI regimen plus bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years
* Histologically confirmed CRC with evidence of metastases and measurable tumor lesions
* Documented disease progression following, or intolerance to, treatment with 5-fluorouracil, oxaliplatin, and bevacizumab-based therapy
* Life expectancy > 3 months
* For patients of reproductive potential (males and females), use of reliable means for contraception (e.g., contraceptive pill, intrauterine device [IUD], physical barrier) throughout the trial and for 6 months following their final exposure to study treatment
* Willingness and capability to be accessible for study follow-up

Exclusion Criteria:

* Patients who have a Kras mutation will be excluded from receiving cetuximab-containing regimens
* Prior radiotherapy to a measurable metastatic lesion(s) to be used for response assessment, unless the lesion has progressed subsequent to the radiotherapy
* Recent radiotherapy to a peripheral lesion, thoracic, abdominal, or pelvic field
* Recent chemotherapy, hormonal therapy, or immunotherapy
* Evidence of clinically detectable ascites
* Other invasive malignancies within 5 years
* History or evidence of active central nervous system (CNS) disease
* Current or recent participation in another experimental drug study
* Clinically significant cardiovascular disease
* Active infection requiring parenteral antibiotics
* Recent major surgical procedure, open biopsy, significant traumatic injury, fine needle aspirations, or anticipation of need for major surgical procedure during the course of the study
* Known or suspected to be positive for the human immunodeficiency virus (HIV)
* Known to be positive for hepatitis C or hepatitis B surface antigen
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or specified study treatment
* Pregnancy (positive pregnancy test) or breast feeding
* Serious, non-healing wound, ulcer, or bone fracture
* Known sensitivity to any of the products administered during the study
* Any disorder that compromises the ability of the patient to provide written informed consent and/or comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities | Through study completion or early study discontinuation

SECONDARY OUTCOMES:
Incidence, nature, and severity of adverse events | Through study completion or early study discontinuation
Change in vital signs | Through study completion or early study discontinuation
Incidence and severity of infusion reactions | Through study completion or early study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Bray, M.D., Study Director — Genentech, Inc.